CLINICAL TRIAL: NCT05766150
Title: Association Between Oral Microbioma With Developing of Oral (Pre)Malignant Disease.
Brief Title: Oral Microbioma and Oral Malignant Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Eliza Hagens, Drs. L.A.A. Vaassen & Dr. E.R.C. Hagens, Academisch Ziekenhuis Maastricht
Other Study IDs: METC 2019-1251
Record Dates: First submitted 2023-02-22; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Oral Cancer; Oral Squamous Cell Carcinoma; Premalignant Lesion
MeSH Terms: conditions — Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with no oral malignant disease
- Patients with oral premalignant disease
- Patients with oral malignant disease

SUMMARY:
This case-control study aims to investigate if oral microbioma is associated with developing oral (pre)malignant disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years in case of oral malignancy or premalignant disease, ≥40 years in case of no malignant disease
* Patients are (partially) dentate (≥20 teeth)
* Patients who have given written informed consent to participate in this study

Exclusion Criteria:

* Patients with a history of radiotherapy in head and neck region
* Patients with a history of chemotherapy, immunotherapy or immunomodulating drugs
* Patients with a previous malginancy in head and neck region
* Edentulous patients (with or without implants)
* Patients with removable (partial) dentures

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Persons visiting oral and maxillofacial surgery department in Maastricht UMC or Radboud UMC who meet the inclusion criteria can be included.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Association between oral microbioma and (pre)malignant disease. | Through study completion, an average of 3 years
  Prevalence of clusters of different oral pathogens will be displayed for patients with malignant disease, premalignant disease and no oral malignancy. Taxonomic representation of statistically and biologically consistent differences between patients with malignant disease, premalignant disease and no oral malignant disease will be displayed.

SECONDARY OUTCOMES:
To describe the difference in oral microbioma between young (>40 years) patients with oral SCC and older (>40 years) patients with oral squamous cell carcinoma. | Through study completion, an average of 3 years
  Prevalence of different oral pathogens will be displayed for patients of both age groups.
To desribe the difference in oral microbioma and stage of disease upon presentation. | Through study completion, an average of 3 years
  Prevalence of different oral pathogens will be displayed for patientgroups with different tumor stages.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Deptartment of Oral and Maxillofacial Surgery, Maastricht UMC+, Maastricht
  - Department of Cranio- & Maxillofacial surgery, Radboud UMC, Nijmegen